CLINICAL TRIAL: NCT06610227
Title: A Clinical Study to Evaluate the Safety, Tolerability, Preliminary Efficacy, and Immunogenicity of the Novel RNA Tumor Vaccine Targeting MICA/B Stress Proteins in Patients With Advanced Solid Tumors
Brief Title: A Study of the RNA Tumor Vaccine Targeting MICA/B in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: NING LI (Other)
Responsible Party: Sponsor-Investigator, NING LI, Director of Clinical Trial Center, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SapRNA-MICA/B
Record Dates: First submitted 2024-09-11; First posted 2024-09-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors
Keywords: RNA vaccine; MICA; MICB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SapRNA™-MICA/B (Experimental): Patients will receive the monotherapy with SapRNA™-MICA/B Tumor Vaccine, which will be administered by intramuscular injection on Day 1, Day 14, and Day 28 respectively.
  Interventions: Biological: SapRNA™-MICA/B Tumor Vaccine

INTERVENTIONS:
Biological: SapRNA™-MICA/B Tumor Vaccine — patients will receive the monotherapy with SapRNA™-MICA/B Tumor Vaccine, which will be administered by intramuscular injection on Day 1, Day 14, and Day 28 respectively

SUMMARY:
This is an open-label, single-arm study to evaluate the safety and efficacy of multiple doses of SapRNA™-MICA/B Tumor Vaccine in patients with advanced solid tumors. Eligible patients will receive the monotherapy with SapRNA™-MICA/B Tumor Vaccine, which will be administered by intramuscular injection on Day 1, Day 14, and Day 28 respectively. Follow-up visits will be performed as scheduled after the end of treatment.

DETAILED DESCRIPTION:
This is an open-label, single-arm study to evaluate the safety and efficacy of multiple doses of SapRNA™-MICA/B Tumor Vaccine in patients with advanced solid tumors. The primary study objective is to evaluate the safety, tolerability, and efficacy of a single dose of SapRNA™-MICA/B Tumor Vaccine in patients. Eligible patients will receive the monotherapy with SapRNA™-MICA/B Tumor Vaccine, which will be administered by intramuscular injection on Day 1, Day 14, and Day 28 respectively. Follow-up visits will be performed as scheduled after the end of treatment. The patients will be followed up until disease progression, occurrence of intolerable toxicity, initiation of a new antitumor therapy, withdrawal of informed consent, loss to follow-up, death, or any other protocol-specified conditions for which the treatment should be discontinued, whichever earlier. Throughout the study, the safety after multiple doses will be evaluated as per the schedule of activities. Endpoints like objective response rate (ORR), disease control rate (DCR), and progression-free survival (PFS) will be evaluated as per the RECIST v1.1 by the investigator. After discontinuation or completion of the study treatment, the end of treatment visit, safety follow-up visit (6 months after end of the last dose), and survival follow-up visit will be performed for the patients.

The dose escalation and tolerability study is proposed to be conducted in the two dose groups of 5×106 and 5×107 active nanoparticles. The patients will receive the treatment at a fixed dose in the study. The dose escalation will be performed with reference to the 3+3 design during the dose-limiting toxicity (DLT) observation period, with 3 patients enrolled first and observed for DLTs from Day 1 to Day 35. If none of the first 3 patients experience DLTs, the study will proceed to the next higher dose level; if 2/3 patients experience DLTs, the study will be stopped; if 1/3 patients experiences DLTs, additional 3 patients will be enrolled: if 1/6 patients experiences DLTs, the study will proceed to the next higher dose level; otherwise, the study will be stopped.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female;
* Expected survival ≥12 weeks;
* Patients with advanced solid tumors as confirmed by cytology or histology who fail standard of care (progressed after treatment or intolerant to the treatment) and have no effective treatment available, or have no standard of care available, or unable to receive standard of care due to limitation of objective conditions;
* Patients with at least 1 measurable lesion as per RECIST v1.1;
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1;
* Patients with adequate organ and bone marrow function. Definitions are as follows:
* Hematology: Absolute neutrophil count (ANC) ≥1.5×109/L; platelet count (PLT) ≥100×109/L; haemoglobin (HGB) ≥9.0 g/dL. No treatment with granulocyte colony stimulating factor (G-CSF), granulocyte macrophage colony stimulating factor (GM-CSF), red blood cell transfusion, and platelet transfusion within 14 days prior to the assessment.
* Liver function:
* Patients with liver metastases: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5×upper limit of normal (ULN), and total bilirubin ≤1.5×ULN (exception: for patients with Gilbert's syndrome, total bilirubin ≤3.0×ULN is acceptable if direct bilirubin ≤35%).
* Patients without liver metastases: AST and ALT ≤2.5×ULN, and total bilirubin ≤1.5×ULN (exception: for patients with Gilbert's syndrome, total bilirubin ≤3.0×ULN is acceptable if direct bilirubin ≤35%).
* Kidney function: Serum creatinine (Scr) ≤1.5×ULN;
* Adequate coagulation function: International normalized ratio (INR) ≤1.5 or prothrombin time (PT) ≤1.5×ULN; it's acceptable to enroll patients who are on anticoagulant therapy as long as the PT is within the established therapeutic range for anticoagulants;
* Left ventricular ejection fraction (LVEF) ≥50% as shown by an echocardiogram (ECHO) or a multigated acquisition (MUGA) scan;
* Willing to sign a written informed consent form and complete the visits and related procedures as required by the protocol.

Exclusion Criteria:

* Patients with autoimmune disease or who are immunosuppressed; requiring treatment with systemic corticosteroids (≥10 mg prednisone, or equivalent dose of other corticosteroids) or immunosuppressants within 14 days prior to the first dose; inhaled and topical steroids are acceptable, or physiological replacement doses of steroids for adrenal insufficiency are acceptable;
* Patients who received major surgery (such as major transabdominal and transthoracic surgeries, excluding diagnostic aspiration or replacement of peripheral intravenous catheters) within 28 days prior to the first dose;
* Patients who received other antitumor therapies within 28 days prior to the first dose or 5 half-lives of the prior antitumor drug (whichever shorter);
* Female patients who are breastfeeding or have positive serum pregnancy test results at screening;
* Patients who experienced any grade 4 immune-related adverse events (irAEs) after receiving prior immunotherapy (patients with endocrine disorders may be enrolled if receiving replacement therapy or experiencing asymptomatic serum amylase and lipase increased), experienced any irAEs leading to permanent discontinuation of treatment after receiving prior immunotherapy, or experienced any grade 3 irAEs within ≤6 months prior to the dose;
* Patients known to have or diagnosed with active central nervous system (CNS) metastases and/or carcinomatous meningitis at screening. However, the following patients may be enrolled: 1) patients with asymptomatic brain metastases (i.e., without progressive CNS symptoms caused by brain metastases, nor requiring treatment with corticosteroids). 2) patients who are treated with stable brain metastases for at least 2 months, without evidence indicating new or enlarged brain metastases;
* Patients with serious cardiovascular and cerebrovascular disorders: inadequately controlled hypertension (systolic blood pressure >160 mmHg, diastolic blood pressure >95 mmHg) after standard of care, symptomatic cardiac insufficiency (NYHA II- IV), unstable angina or myocardial infarction within 6 months, or patients with risks of QTc interval prolongation or arrhythmia (QTcF >470 ms at baseline, uncorrected hypokalaemia, long QT syndrome, atrial fibrillation with heart rate >100 bpm at rest, or serious cardiac valve disease);
* Patients with uncontrolled pleural effusion, ascites, and pericardial effusion;
* Patients with active infections requiring treatment: active Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection; known history of human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS); active tuberculosis, etc.;
* Patients with toxicities from prior antitumor therapies which fail to return to CTCAE grade ≤1 (NCI-CTCAE v5.0) or baseline level, excluding atrichia and skin pigmentation (any grades);
* Patients with a history of severe allergic reactions to biologics;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
adverse events | From enrollment to the end of treatment at 30 days
  Frequency, number, incidence, and severity of the adverse events and adverse reactions

SECONDARY OUTCOMES:
Objective response rate (ORR) | Every 6 weeks from the first dose of treatment until the date of first documented progression, the start of other treatment, or date of death from any cause, whichever came first, up to 2 years
  Objective response rate will be estimated by CT or MRI depending on the cancer type and location, according to RESIST V1.1.
Immunogenicity | 1 hour before injection at Day 1, Day 14, and Day 28, and then Week 7 and Week 16
  Change in vaccine-specific antibody (IgG) after treatment will be measured.
Target protein expression | 1 hour before injection at Day 1, and then Week 7 and Week 16
  Levels of serum MICA/B stress proteins will be measured by ELISA.

OTHER OUTCOMES:
MICA/B-specific CD4+ and CD8+ T lymphocytes | 1 hour before injection at Day 1, and then Week 7 and Week 16
  Responses of antigen-specific CD4+ and CD8+ T lymphocytes after treatment with SapRNA™-MICA/B Tumor Vaccine. ELISPOT will be used for detection of antigen-specific CD4+ and CD8+ T lymphocytes.
NK cells in peripheral blood | 1 hour before injection at Day 1, and then Week 7 and Week 16
  Responses of natural killer (NK) cells after treatment with SapRNA™-MICA/B Tumor Vaccine. Flow cytometry will be used for NK cell measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, M.D., Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The decision will be made after completion of this study.